CLINICAL TRIAL: NCT03376607
Title: Community- and mHealth-Based Integrated Management of Diabetes in Primary Healthcare in Rwanda: The D²Rwanda Study
Brief Title: Community- and mHealth-Based Integrated Management of Diabetes in Primary Healthcare in Rwanda
Acronym: D²Rwanda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Luxembourg (Other); Karen Elise Jensens Fond (Unknown); University of Rwanda (Other); Rwanda Biomedical Centre (Other); Luxembourg Institute of Socio-Economic Research (LISER) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D²Rwanda
Record Dates: First submitted 2017-12-06; First posted 2017-12-18 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Telemedicine; Community Health Workers
Keywords: Primary Health Care; Health Behavior; Quality of Life; Health Literacy; Global Health; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): Intervention group 1 will receive access to the newly-established HBCP programme.
  Interventions: Other: HBCP programme
- Intervention group 2 (Experimental): Intervention group 2 will receive access to the newly-established HBCP programme, and facilitated access to a mobile health application.
  Interventions: Other: HBCP programme; Behavioral: mobile health application
- Control group (No Intervention): The control group will receive routine practice.

INTERVENTIONS:
Other: HBCP programme — The newly-established Home-Based Community Practitioners (HBCPs) programme will enable frontline workers to offer monthly health assessments, disease management and lifestyle advice to diabetic patients, and referral to the district hospitals when needed.
  Other Names: Intervention 1
  Arms: Intervention group 1; Intervention group 2
Behavioral: mobile health application — HBCPs will actively encourage the use of a mobile app by assisting patients to access it (this process is known as "facilitated access"). The app will enable: (i) the registration of measurements, such as blood glucose and weight; (ii) the registration of concerns and questions in a diary; (iii) the reception of alerts and notifications for the appointments to the health facilities, and; (iv) access to advice on lifestyle improvement and other patient educational material.
  Other Names: Intervention 2
  Arms: Intervention group 2

SUMMARY:
The Home Based Care Practitioners (HBCPs) programme has been established by the Rwandan Ministry of Health in response to the shortage of health professionals. Currently in its pilot first phase, it entails laypeople providing longitudinal care to chronic patients after receiving a six-month training.The diabetes mellitus (DM) prevalence in Rwanda is estimated at 3.5%. Technological mobile solutions can improve care by enabling patients to self-manage their disease.

It is hypothesised that the establishment of the HBCP programme with regular monthly assessments of DM patients and disease management by the programme's HBCPs improves the patients' HbA1c levels, medication adherence, health-related quality of life, mental well-being, and health literacy levels. It is also hypothesised that patients will show further improvement when the HBCP programme is coupled with a mobile health application for patients that includes diaries, notifications and educational material. The aim of the study is to determine the efficacy of such an integrated programme for the management of DM in primary health care in Rwanda.

Study design: The study is designed as a one-year, open-label cluster trial of two interventions (intervention 1: HBCP programme; intervention 2: HBCP programme + mobile health application) and usual care (control). In preparation for the onset of the study, a mobile application is being developed. Focus discussion groups will be carried out with selected patients and HBCPs after the end of the main trial to explore their opinions in participating in the study.

Study population: District hospitals from those running the HBCP programme will be selected according to criteria. Under each district hospital, the administrative areas ("cells") participating in the HBCP programme will be randomised to receive intervention 1 or 2. The patients from each group who meet the eligibility criteria of the study will receive the same intervention. Cells that do not participate in HBCP programme will be assigned to the control group.

Study endpoints: The primary outcomes will be changes in HbA1c levels. Medication adherence, mortality, complications, health-related quality of life, mental well-being and health literacy will be assessed as secondary outcomes.

Sponsor: The D²Rwanda project has received financial support by the Karen Elise Jensens Fond (Denmark), and the Universities of Aarhus and Luxembourg.

DETAILED DESCRIPTION:
Background: In Rwanda, diabetes mellitus (DM) prevalence has been estimated between 3.0 - 3.5%. Several factors, including an increase in screening and diagnosis programmes, the urbanization of the population, and changes in lifestyle are likely to contribute to a sharp increase in the prevalence of DM in the next decade, posing a daunting challenge for the fragile health care systems in low- and middle-income countries (LMICs). At the same time, the level of knowledge and perceptions of DM among patients is inadequate. Patients with low health literacy levels are often unable to recognise the signs and symptoms of DM, and may access their health provider late, hence presenting with more complications.

Although the majority of the Rwandan population seek care at the health centres, the Rwandan primary health care is facing a shortage of human resources. A community health worker programme was introduced in Rwanda in 2007 covering mainly infectious diseases, maternal and child health, and family planning.

In response to the need for better management of non-communicable diseases (NCDs) at the community level, the Ministry of Health of Rwanda and its partners adopted a new strategy and initiated a Home-Based Care Practitioner (HBCP) programme. Approximately 100 cells, belonging to the catchment area of nine selected hospitals, participate in the first phase of the HBCP programme (a "cell" is a small administrative area under the larger areas called "districts"). Every cell has two HBCPs, who completed high school and received six months of technical vocational education and training organised by the Ministry of Health in collaboration with its partners.

There is growing evidence for the efficacy of interventions using mobile devices (mHealth) in LMICs, particularly in improving treatment adherence, appointment compliance, data gathering, and developing support networks for health workers. In Rwanda, there is an urgent call to using mHealth interventions for the prevention and management of NCDs. The present research project responds to this by developing an mHealth intervention integrated in the current primary health care system, in support of both the DM patients and their healthcare providers.

Randomisation: The unit of randomisation will be the cluster, defined by the cell. In each cell two HBCPs work. Under each district hospital, the cells participating in the HBCP programme will be randomised to receive intervention 1 or 2. The patients from each group will receive the same intervention. An equal number of cells, out of those not participating in the HBCP programme, will be randomly selected and assigned to the control group.

Sample size: Lacking other data on diabetes in Rwanda, the standard deviation from a study of Levitt et al. in South Africa is used to calculate the within and between variance. A one-point difference in HbA1c is considered as clinically significant outcome based on previous studies. For the power calculation, a within variance of 4.76, a between variance of 0.53, and an intra-class correlation of 0.1 are assumed. Based on the information which will be gathered before the onset of the trial, the final sample will be estimated assuming either four or six patients per cell (in each cell two HBCPs work).

Assuming four patients per cell, the number of clusters per group needed is 27 for a total number of 108 patients per group to achieve 80% power with a 5% level of significance (total number of patients: 324, total number of cells: 81). 144 patients per group (total number of patients: 432; total number of cells: 108) will be needed to allow for a 30% attrition.

Assuming six patients per cell, the number of clusters per group needed is 21 for a total number of 126 patients per group to achieve 80% power with a 5% level of significance (total number of patients: 378, total number of cells: 63). 168 patients per group (total number of patients: 504; total number of cells: 84) will be needed to allow for a 30% attrition.

Study questionnaires: Four questionnaires will be employed for the assessment of the patients of the trial (D-39, PAID, BMQ, ISHA-Q). In preparation for their use both their translation in Kinyarwanda and their cultural adaptation will be carried out.

Qualitative study: At the end of the trial two types of focus discussion groups will be conducted: a) with patients of the two intervention groups, and; b) with HBCPs delivering the two interventions of the study. The aim of these focus discussion groups is to explore the ways the intervention will have been enacted in practice, expected and unexpected impacts, and the perceptions of relevance and contextual issues that may have impacted the intervention.

Ethical review: Ethical approval has been obtained from the Rwanda National Ethics Committee (100/RNEC/2017; amendment approved in 463/RNEC/2017; renewed in 113/RNEC/2018) and the Ethics Review Panel of the University of Luxembourg (ERP 17-014 D2Rwanda; amendment approved in ERP 17-048 D2Rwanda).

ELIGIBILITY:
Inclusion Criteria for patients:

1. Adult patients (male and female) aged between 21 and 80 years
2. Diagnosed and confirmed as diabetic patient at least 6 months prior to study start
3. Living in the administrative areas (called "cells") of the district hospitals participating in the first phase of the HBCP programme
4. Residing, and planning to reside within a 2-hour travel distance on foot from the study site for the duration of follow-up
5. Willing and able to adhere to the study protocol
6. Willing and able to give informed consent for enrolment in the study

Exclusion Criteria for patients:

1. Severe mental health conditions, including cognitive impairments, as registered in their clinical records
2. Severe hearing and visual impairments as registered in their clinical records
3. Terminal illness
4. Illiteracy
5. Pregnancy or post-partum period

Inclusion criteria for HBCPs:

1. Permanent residence in one of the cells of the study
2. Willing and able to give informed consent for enrolment in the study

Exclusion criteria for HBCPs:

1. Not capable of accomplishing questionnaires due to reading or communication problems

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Change from baseline to 12-month follow-up

SECONDARY OUTCOMES:
Change in medication adherence | Change from baseline to 6- and 12-month follow-up
  To assess medication adherence and evaluate patients' medication-taking behaviour, reported side-effects, concerns and barriers to adherence, the Kinyarwanda version of the Brief Medication Questionnaire (BMQ) will be administered at: baseline, after six months, and on trial completion (after 12 months). Data will also be gathered from the pharmacies dispensing medications to calculate the pill count, in an attempt to triangulate the information received from the BMQ with a more objective method.
Number of dropouts of the NCD clinics of the district hospitals | From baseline to 12-month follow-up
Number of lost appointments to the NCD clinics of the district hospitals | From baseline to 12-month follow-up
Mortality | From baseline to 12-month follow-up
Number of complications | From baseline to 12-month follow-up
Number of referrals | From baseline to 12-month follow-up
Change in health literacy | Change from baseline to 12-month follow-up
  The Kinyarwanda version of the Information and Support for Health Actions Questionnaire (ISHA-Q) will be employed to assess the health literacy level (at baseline and after 12 months).
Change in health-related quality of life | Change from baseline to 6- and 12-month follow-up
  The Kinyarwanda version of the Diabetes-39 (D-39) questionnaire will be used to measure health-related quality of life (at baseline, after six months, and on trial completion (after 12 months)).
Change in mental well-being | Change from baseline to 6- and 12-month follow-up
  The Kinyarwanda version of the Problem Areas in Diabetes questionnaire (PAID) questionnaire will be administered to evaluate psychological well-being (at baseline, after six months, and on trial completion (after 12 months)).
Percentage of patients with at least one measurement of HbA1c | Change from baseline to 12-month follow-up
Percentage of patients with at least one measurement of fasting blood glucose (FBG) levels | Change from baseline to 12-month follow-up
Percentage of patients with at least one measurement of creatinine | Change from baseline to 12-month follow-up
Percentage of patients with at least one measurement of urine proteins (dipstick) | Change from baseline to 12-month follow-up
Percentage of patients with at least one measurement of blood pressure | Change from baseline to 12-month follow-up
Percentage of patients with at least one recording of body mass index (BMI) | Change from baseline to 12-month follow-up
Fasting blood glucose (FBG) | Change from baseline to 12-month follow-up
Creatinine | Change from baseline to 12-month follow-up
Urine proteins (dipstick) | Change from baseline to 12-month follow-up
Blood pressure | Change from baseline to 12-month follow-up
Body mass index (BMI) | Change from baseline to 12-month follow-up
Recorded number of smokers | Change from baseline to 12-month follow-up
  Recording of whether a patient is smoker or not
Number of patients with recorded pack years | Change from baseline to 12-month follow-up
  Pack years are calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked
Number of patients with recorded alcohol intake per week | Change from baseline to 12-month follow-up
Number of smokers | Change from baseline to 12-month follow-up
Number of cigarettes per day | Change from baseline to 12-month follow-up
Alcohol intake per week | Change from baseline to 12-month follow-up

OTHER OUTCOMES:
Patients' challenges receiving care | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
Patients understanding of diabetes' natural history | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
How the patients' disease-related decision-making is influence | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
How the patients' disease-related decision-making is influenced | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
The challenges of patients in using the mobile app | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
The changes in behaviour that the intervention brought about | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with patients
The challenges in the work of HBCPs | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with HBCPs
The level of satisfaction of HBCPs | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with HBCPs
The challenges in integrating the app to the usual visits | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with HBCPs
The differences the HBCPs note from patient to patient | On trial completion (approximately after 12 months)
  The qualitative part of the study will include focus discussion groups and interviews with HBCPs

CONTACTS AND LOCATIONS:
Overall Officials: Per Kallestrup, MD, PhD, Principal Investigator — University of Aarhus; Claus Vögele, DPsych, PhD, Principal Investigator — University of Luxembourg; Jeanine Condo Umutesi, MD, MSc, PhD, Principal Investigator — Rwanda Biomedical Centre; Conchitta D'Ambrosio, MSc, PhD, Principal Investigator — University of Luxembourg
Locations (9):
- Rwanda (9):
  - Kibuye Referral Hospital, Kibuye, Karongi
  - Ruhengeri Provincial Hospital, Ruhengeri, Musanze
  - Kibungo Referral Hospital, Kibungo, Ngoma
  - Bushenge Provincial Hospital, Bushenge, Nyamasheke
  - Muhima District Hospital, Kigali, Nyarugenge
  - Ruhango Provincial Hospital, Kinazi, Ruhango
  - Kinihira Provincial Hospital, Kinihira, Rulindo
  - Kabutare District Hospital, Huye
  - Rwamagana Provincial Hospital, Rwamagana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] World Health Organization (WHO). Global status report on noncommunicable diseases 2014. 2014;298. Available from: http://www.who.int/nmh/publications/ncd-status-report-2014/en/
- [Background] Hilawe EH, Yatsuya H, Kawaguchi L, Aoyama A. Differences by sex in the prevalence of diabetes mellitus, impaired fasting glycaemia and impaired glucose tolerance in sub-Saharan Africa: a systematic review and meta-analysis. Bull World Health Organ. 2013 Sep 1;91(9):671-682D. doi: 10.2471/BLT.12.113415. PMID 24101783
- [Background] Tapela N, Habineza H, Anoke S, Harerimana E, Mutabazi F, Hedt-Gauthier B, et al. Diabetes in Rural Rwanda: High Retention and Positive Outcomes after 24 Months of Follow-up in the Setting of Chronic Care Integration. Int J Diabetes Clin Res [Internet]. 2016 [cited 2016 Dec 5];3(2). Available from: http://clinmedjournals.org/articles/ijdcr/international-journal-of-diabetes-and-clinical-research-ijdcr-3-058.php
- [Background] Hall V, Thomsen RW, Henriksen O, Lohse N. Diabetes in Sub Saharan Africa 1999-2011: epidemiology and public health implications. A systematic review. BMC Public Health. 2011 Jul 14;11:564. doi: 10.1186/1471-2458-11-564. PMID 21756350
- [Background] World Health Organization (WHO). WHO STEPwise approach to Surveillance (STEPS). 2013.
- [Background] International Diabetes Federation (IDF). IDF Diabetes Atlas 7th edition [Internet]. idf.org. Brussels; 2015. Available from: http://www.diabetesatlas.org/
- [Background] Windus DW, Ladenson JH, Merrins CK, Seyoum M, Windus D, Morin S, Tewelde B, Parvin CA, Scott MG, Goldfeder J. Impact of a multidisciplinary intervention for diabetes in Eritrea. Clin Chem. 2007 Nov;53(11):1954-9. doi: 10.1373/clinchem.2007.095067. PMID 17954497
- [Background] Mukeshimana MM, Nkosi ZZ. Communities' knowledge and perceptions of type two diabetes mellitus in Rwanda: a questionnaire survey. J Clin Nurs. 2014 Feb;23(3-4):541-9. doi: 10.1111/jocn.12199. Epub 2013 Jun 21. PMID 23789978
- [Background] Schillinger D, Grumbach K, Piette J, Wang F, Osmond D, Daher C, Palacios J, Sullivan GD, Bindman AB. Association of health literacy with diabetes outcomes. JAMA. 2002 Jul 24-31;288(4):475-82. doi: 10.1001/jama.288.4.475. PMID 12132978
- [Background] Gill GV, Mbanya JC, Ramaiya KL, Tesfaye S. A sub-Saharan African perspective of diabetes. Diabetologia. 2009 Jan;52(1):8-16. doi: 10.1007/s00125-008-1167-9. Epub 2008 Oct 10. PMID 18846363
- [Background] National Institute of Statistics of Rwanda. Rwanda Integrated Household Living Conditions Survey (EICV) 2013/2014. 2014.
- [Background] National Institute of Statistics of Rwanda (NISR). The Statistical Yearbook, 2014 Edition [Internet]. 2014. Available from: http://statistics.gov.rw/publications/statistical-yearbook-2014
- [Background] Ministry of Health (MOH) [Rwanda]. Non communicable diseases policy [Internet]. 2015. Available from: http://www.moh.gov.rw/fileadmin/templates/policies/NCDs_Policy.2015.pdf
- [Background] National Institute of Statistics of Rwanda. Statistical Yearbook 2014. 2014.
- [Background] Campbell J, Buchan J, Cometto G, David B, Dussault G, Fogstad H, Fronteira I, Lozano R, Nyonator F, Pablos-Mendez A, Quain EE, Starrs A, Tangcharoensathien V. Human resources for health and universal health coverage: fostering equity and effective coverage. Bull World Health Organ. 2013 Nov 1;91(11):853-63. doi: 10.2471/BLT.13.118729. PMID 24347710
- [Background] Ministry of Health (MOH) [Rwanda]. Health Sector Policy [Internet]. Kigali; 2014. Available from: http://www.moh.gov.rw/fileadmin/templates/policies/Health_Sector_Policy_2014.pdf
- [Background] Fox LM, Ravishankar N, Squires J, Williamson RT, Derick B. Rwanda Health Governance Report [Internet]. Bethesda, MD; 2010. Available from: http://apps.who.int/medicinedocs/documents/s18413en/s18413en.pdf
- [Background] Agarwal S, Rosenblum L, Goldschmidt T, Carras M, Goal N, Labrique AB. Mobile Technology in Support of Frontline Health Workers. John Hopkins Univ Glob mHealth Initiat 2016 [Internet]. 2016;86. Available from: https://dl.dropboxusercontent.com/u/5243748/mFHW Landscape_2016 Final.pdf
- [Background] Braun R, Catalani C, Wimbush J, Israelski D. Community health workers and mobile technology: a systematic review of the literature. PLoS One. 2013 Jun 12;8(6):e65772. doi: 10.1371/journal.pone.0065772. Print 2013. PMID 23776544
- [Background] Binagwaho A. Role of community health in strengthening Rwandan health system [Internet]. 2011 [cited 2016 Feb 6]. Available from: http://www.webcitation.org/6f5urhqiP
- [Background] Condo J, Mugeni C, Naughton B, Hall K, Tuazon MA, Omwega A, Nwaigwe F, Drobac P, Hyder Z, Ngabo F, Binagwaho A. Rwanda's evolving community health worker system: a qualitative assessment of client and provider perspectives. Hum Resour Health. 2014 Dec 13;12:71. doi: 10.1186/1478-4491-12-71. PMID 25495237
- [Background] Farmer PE, Nutt CT, Wagner CM, Sekabaraga C, Nuthulaganti T, Weigel JL, Farmer DB, Habinshuti A, Mugeni SD, Karasi JC, Drobac PC. Reduced premature mortality in Rwanda: lessons from success. BMJ. 2013 Jan 18;346:f65. doi: 10.1136/bmj.f65. PMID 23335479
- [Background] Joshi R, Alim M, Kengne AP, Jan S, Maulik PK, Peiris D, Patel AA. Task shifting for non-communicable disease management in low and middle income countries--a systematic review. PLoS One. 2014 Aug 14;9(8):e103754. doi: 10.1371/journal.pone.0103754. eCollection 2014. PMID 25121789
- [Background] Mishra SR, Neupane D, Preen D, Kallestrup P, Perry HB. Mitigation of non-communicable diseases in developing countries with community health workers. Global Health. 2015 Nov 10;11:43. doi: 10.1186/s12992-015-0129-5. PMID 26555199
- [Background] Kok MC, Dieleman M, Taegtmeyer M, Broerse JE, Kane SS, Ormel H, Tijm MM, de Koning KA. Which intervention design factors influence performance of community health workers in low- and middle-income countries? A systematic review. Health Policy Plan. 2015 Nov;30(9):1207-27. doi: 10.1093/heapol/czu126. Epub 2014 Dec 11. PMID 25500559
- [Background] Hill Z, Dumbaugh M, Benton L, Kallander K, Strachan D, ten Asbroek A, Tibenderana J, Kirkwood B, Meek S. Supervising community health workers in low-income countries--a review of impact and implementation issues. Glob Health Action. 2014 May 8;7:24085. doi: 10.3402/gha.v7.24085. eCollection 2014. PMID 24815075
- [Background] United Nations Economic and Social Commission for Asia and the Pacific 2017. Bloomberg Data for Health Initiative. 201.
- [Background] Ministry of Health (MOH) [Rwanda]. Health Sector Annual Report: July 2015-June 2016 [Internet]. Kigali; 2016. Available from: http://www.moh.gov.rw/fileadmin/templates/MOH-Reports/Health_20Sector_20Annual_20Report_202015-2016_25082016.pdf
- [Background] Stephani V, Opoku D, Quentin W. A systematic review of randomized controlled trials of mHealth interventions against non-communicable diseases in developing countries. BMC Public Health. 2016 Jul 15;16:572. doi: 10.1186/s12889-016-3226-3. PMID 27417513
- [Background] Vital Wave Consulting. mHealth for Development: The Opportunity of Mobile Technology for Healthcare in the Developing World [Internet]. Washington, D.C.; 2009. Available from: http://www.unfoundation.org/what-we-do/issues/global-health/mhealth-report.html
- [Background] GSMA. The Mobile Economy: Sub Saharan Africa 2014 [Internet]. London, United Kingdom; 2014. Available from: http://www.gsmamobileeconomyafrica.com/GSMA_ME_SubSaharanAfrica_Web_Singles.pdf
- [Background] National Institute of Statistics of Rwanda (NISR) [Rwanda], Ministry of Health (MOH) [Rwanda], ICF International. Rwanda Demographic and Health Survey 2014-15. Rockville, Maryland, USA: NISR, MOH, and ICF International; 2015.
- [Background] Utilities Rwanda Regulatory Authority. Statistics and tariff information in telecommunication, media and postal service as of the fourth quarter 2016 [Internet]. 2016. Available from: http://www.rura.rw/fileadmin/docs/statistics/Statistics_report_4th_quarter___2016_for_publication_.pdf
- [Background] World Health Organization (WHO). ITU and WHO launch mHealth initiative to combat noncommunicable diseases [Internet]. 2012 [cited 2016 Feb 6]. Available from: http://www.who.int/nmh/events/2012/mhealth/en/
- [Background] Bloomfield GS, Vedanthan R, Vasudevan L, Kithei A, Were M, Velazquez EJ. Mobile health for non-communicable diseases in Sub-Saharan Africa: a systematic review of the literature and strategic framework for research. Global Health. 2014 Jun 13;10:49. doi: 10.1186/1744-8603-10-49. PMID 24927745
- [Background] Asiimwe-kateera B, Condo J, Ndagijimana A, Kumar S, Mukeshimana M, Gaju E, et al. Mobile Health Approaches to Non-Communicable Diseases in Rwanda. 2015;2(1):89-92.
- [Background] Torjesen I. Maternal deaths have nearly halved in past 25 years. BMJ. 2015 Nov 13;351:h6129. doi: 10.1136/bmj.h6129. No abstract available. PMID 26566922
- [Background] International Diabetes Federation. Global Diabetes Scorecard Tracking Progress for Action [Internet]. Bruxelles; 2014. Available from: http://www.idf.org/global-diabetes-scorecard/assets/downloads/Scorecard-29-07-14.pdf
- [Background] World Health Organization (WHO). Adherence to long-term therapies: evidence for action. 2003;2014:1-194. Available from: http://www.who.int/chp/knowledge/publications/adherence_full_report.pdf
- [Background] Bagonza J, Rutebemberwa E, Bazeyo W. Adherence to anti diabetic medication among patients with diabetes in eastern Uganda; a cross sectional study. BMC Health Serv Res. 2015 Apr 19;15:168. doi: 10.1186/s12913-015-0820-5. PMID 25898973
- [Background] Cramer JA. A systematic review of adherence with medications for diabetes. Diabetes Care. 2004 May;27(5):1218-24. doi: 10.2337/diacare.27.5.1218. PMID 15111553
- [Background] Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24;17(2):e52. doi: 10.2196/jmir.3951. PMID 25803266
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Torgerson DJ. Contamination in trials: is cluster randomisation the answer? BMJ. 2001 Feb 10;322(7282):355-7. doi: 10.1136/bmj.322.7282.355. No abstract available. PMID 11159665
- [Background] Lopez-Pelayo H, Wallace P, Segura L, Miquel L, Diaz E, Teixido L, Baena B, Struzzo P, Palacio-Vieira J, Casajuana C, Colom J, Gual A. A randomised controlled non-inferiority trial of primary care-based facilitated access to an alcohol reduction website (EFAR Spain): the study protocol. BMJ Open. 2014 Dec 31;4(12):e007130. doi: 10.1136/bmjopen-2014-007130. PMID 25552616
- [Background] Boyer JG, Earp JA. The development of an instrument for assessing the quality of life of people with diabetes. Diabetes-39. Med Care. 1997 May;35(5):440-53. doi: 10.1097/00005650-199705000-00003. PMID 9140334
- [Background] Garratt AM, Schmidt L, Fitzpatrick R. Patient-assessed health outcome measures for diabetes: a structured review. Diabet Med. 2002 Jan;19(1):1-11. doi: 10.1046/j.1464-5491.2002.00650.x. PMID 11869297
- [Background] Watkins K, Connell CM. Measurement of health-related QOL in diabetes mellitus. Pharmacoeconomics. 2004;22(17):1109-26. doi: 10.2165/00019053-200422170-00002. PMID 15612830
- [Background] Speight J, Reaney MD, Barnard KD. Not all roads lead to Rome-a review of quality of life measurement in adults with diabetes. Diabet Med. 2009 Apr;26(4):315-27. doi: 10.1111/j.1464-5491.2009.02682.x. PMID 19388959
- [Background] Dodson S, Good S, Osborne R. Health literacy toolkit for low- and middle-income countries: a series of information sheets to empower communities and strengthen health systems [Internet]. National Network of Libraries of Medicine Southeastern/Atlantic Region. New Delhi: World Health Organization, Regional Office for South-East Asia; 2015. Available from: http://apps.searo.who.int/PDS_DOCS/B5148.pdf?ua=1
- [Background] Svarstad BL, Chewning BA, Sleath BL, Claesson C. The Brief Medication Questionnaire: a tool for screening patient adherence and barriers to adherence. Patient Educ Couns. 1999 Jun;37(2):113-24. doi: 10.1016/s0738-3991(98)00107-4. PMID 14528539
- [Background] Lavsa SM, Holzworth A, Ansani NT. Selection of a validated scale for measuring medication adherence. J Am Pharm Assoc (2003). 2011 Jan-Feb;51(1):90-4. doi: 10.1331/JAPhA.2011.09154. PMID 21247831
- [Background] Lam WY, Fresco P. Medication Adherence Measures: An Overview. Biomed Res Int. 2015;2015:217047. doi: 10.1155/2015/217047. Epub 2015 Oct 11. PMID 26539470
- [Background] Levitt NS, Bradshaw D, Zwarenstein MF, Bawa AA, Maphumolo S. Audit of public sector primary diabetes care in Cape Town, South Africa: high prevalence of complications, uncontrolled hyperglycaemia, and hypertension. Diabet Med. 1997 Dec;14(12):1073-7. doi: 10.1002/(SICI)1096-9136(199712)14:123.0.CO;2-9. PMID 9455936
- [Background] Mash RJ, Rhode H, Zwarenstein M, Rollnick S, Lombard C, Steyn K, Levitt N. Effectiveness of a group diabetes education programme in under-served communities in South Africa: a pragmatic cluster randomized controlled trial. Diabet Med. 2014 Aug;31(8):987-93. doi: 10.1111/dme.12475. Epub 2014 May 20. PMID 24766179
- [Background] van Teijlingen E, Hundley V. The importance of pilot studies. Nurs Stand. 2002 Jun 19-25;16(40):33-6. doi: 10.7748/ns2002.06.16.40.33.c3214. PMID 12216297
- [Background] Schenker MB, Castañeda X, Rodriguez-Lainz A, editors. Migration and Health - A Research Methods Handbook. Oakland, California: University of California Press; 2014
- [Background] Mrc, Clark A, Clark A. Anonymising Research Data. Sociol J Br Sociol Assoc. 2006;44:1-48
- [Derived] Lygidakis C, Uwizihiwe JP, Bia M, Uwinkindi F, Kallestrup P, Vogele C. Quality of life among adult patients living with diabetes in Rwanda: a cross-sectional study in outpatient clinics. BMJ Open. 2021 Feb 19;11(2):e043997. doi: 10.1136/bmjopen-2020-043997. PMID 33608403
- [Derived] Lygidakis C, Uwizihiwe JP, Kallestrup P, Bia M, Condo J, Vogele C. Community- and mHealth-based integrated management of diabetes in primary healthcare in Rwanda (D(2)Rwanda): the protocol of a mixed-methods study including a cluster randomised controlled trial. BMJ Open. 2019 Jul 24;9(7):e028427. doi: 10.1136/bmjopen-2018-028427. PMID 31345971
- See also: Karen Elise Jensens Fond is the main sponsor of the study — http://www.kejfond.dk